CLINICAL TRIAL: NCT02762877
Title: A Study to Determine the Concordance of Key Actionable Genomic Alterations as Assessed in Tumor Tissue and Plasma From Patients With Non Small Cell Lung Carcinoma (NSCLC)
Brief Title: Concordance of Key Actionable Genomic Alterations as Assessed in Tumor Tissue and Plasma in Non Small Cell Lung Cancer
Status: Terminated | Type: Observational
Why Stopped: Business decision
Sponsor: Genomic Health®, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 14-009
Record Dates: First submitted 2016-04-29; First posted 2016-05-05 (Estimated); Results first posted 2019-11-25 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Non Small Cell Lung Carcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and tissue

GROUPS / COHORTS (2):
- A: Patients with non-squamous NSCLC either newly diagnosed or progressing on any therapy (except erlotinib, gefitinib, or afatinib)
- B: Patients with non-squamous NSCLC who are progressing on erlotinib, gefitinib, or afatinib

SUMMARY:
A study to determine the concordance of key actionable genomic alterations as assessed in tumor tissue and plasma from patients with non small cell lung carcinoma (NSCLC)

DETAILED DESCRIPTION:
This is a prospective clinical study to characterize the concordance of key clinically relevant genomic alterations in tumor tissue (biopsy/excision/cytology) and liquid biopsy (blood) using the Genomic Health LBMP in patients with stage IV non squamous NSCLC, that are either newly diagnosed with metastatic disease or progressing on therapy (any line). Tissue biopsy and blood collection (liquid biopsy) should be less than eight weeks apart and with no new systemic antitumoral treatment given in the interval between the tissue biopsy and blood collection. Local assessment of tumor tissue samples will be performed at each participating institution as per their clinical standard of care practices and results from the local assessment of genomic alteration status will be used.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be 18 years or older.
* Patients with stage IV non squamous NSCLC who are either newly diagnosed or progressing on any treatment (progression defined as increasing tumor size or new metastatic lesions on clinical or imaging assessment).
* Patients with available tissue sample from a metastatic site or, if the patient presents with stage IV disease at diagnosis, from the primary tumor or a metastatic site. If a patient is progressing on EGFR targeted therapy (erlotinib, gefitinib, afatinib), tumor tissue sample is required only if available.
* No new systemic anti-tumor therapy administered in the interval between the tissue biopsy and collection of the blood sample. (interval not to exceed eight weeks). Local radiation therapy is permitted.
* Able and willing to read, understand and sign an informed consent and Health Insurance Portability and Accountability Act (HIPAA) authorization, or equivalent privacy law, where this is applicable.

Exclusion Criteria:

* Patients who are currently receiving therapy (targeted, immune- or chemotherapy) without sign of progression.
* Patients with squamous NSCLC.
* Patients with more than 8 weeks between collection of tumor specimen and collection of blood sample for analysis. (Not applicable for patients progressing on EGFR targeted therapy with no biopsy at progression)
* Patients changing EGFR therapy due to toxicity or preference without documented disease progression.
* Patients progressing on Osimertinib treatment.
* Patients with brain metastases only.
* Inability to comply with study and/or follow-up procedures.
* Unable or unwilling to provide written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Non small cell lung cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2016-04; Primary Completion 2018-07-01 (Actual); Study Completion 2019-06-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (22):
- United States (9):
  - Cancer Care Associates d/b/a Torrance Memorial Physician Network, Torrance, California
  - Central Georgia Cancer Care, Macon, Georgia
  - Virginia Piper Cancer Institute, Minneapolis, Minnesota
  - Essex Oncology of North Jersey, Belleville, New Jersey
  - Meridian Hospitals, Neptune City, New Jersey
  - Gabrail Cancer Center, Canton, Ohio
  - West Clinic, Germantown, Tennessee
  - Bon Secours Cancer Institute, Midlothian, Virginia
  - MultiCare Health System, Tacoma, Washington
- Chile (3):
  - Instituto Nacional del Torax, Santiago
  - Fundación Arturo López Perez, Santiago
  - Clinica Alemana de Santiago, Santiago
- France (3):
  - Centre Jean Perrin, Clermont-Ferrand, Cedex 1
  - Hôpital Nord, Marseille, Cedex 20
  - Polyclinique Bordeaux Nord Aquitaine, Bordeaux
- St. Vincent's University Hospital, Dublin, Elm Park, Ireland
- Japan (2):
  - Tokyo Medical University Hospital, Tokyo, Shinjuku-ku
  - National Cancer Center, Tokyo, Tsukiji, Chuo-ku
- Spain (3):
  - Hospital Universitario Central Asturias, Oviedo
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Clinico Universitario Lozano Blesa, Zaragoza
- Clatterbridge Cancer Center NHS Foundation Trust, Bebington, Wirral, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- A - NSCLC All Comers Regardless of Genomic Alteration Status: Patients with non-squamous NSCLC regardless of genomic alteration status (newly diagnosed or progressing on therapy)
- B - Progressing on EGFR Targeted Therapies: Patients with non-squamous NSCLC progressing on erlotinib, gefitinib, or afatinib
Period: Overall Study
Arm/Group | A - NSCLC All Comers Regardless of Genomic Alteration Status | B - Progressing on EGFR Targeted Therapies
Started | 121 | 19
Completed | 121 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | A - NSCLC All Comers Regardless of Genomic Alteration Status | B - Progressing on EGFR Targeted Therapies | Total
Number analyzed (Participants) | 121 | 19 | 140
Age, Customized [Median (Full Range); unit: years]
  Age, years | 66 [42 to 94] | 67 [45 to 85] | 66 [42 to 94]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 10 | 71
  Male | 60 | 9 | 69
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 91 | 12 | 103
  Not Hispanic or Latino | 3 | 1 | 4
  Unknown or Not Reported | 27 | 6 | 33
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 14 | 4 | 18
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 0 | 8
  White | 74 | 9 | 83
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 25 | 6 | 31
EGFR Mutation Tested [Count of Participants; unit: Participants] — Patients who received EGFR mutation testing on both their tissue and plasma samples.
  Participants | 117 | 19 | 136
ALK-EML4 Fusion Mutation Tested [Count of Participants; unit: Participants] — Patients who received ALK (EML4-ALK fusion) mutation testing on both their tissue and plasma samples.
  Participants | 115 | NA — Patients enrolled in Arm B were only assessed for EGFR mutation testing. | NA — Total not calculated because data are not available (NA) in one or more arms.

OUTCOME MEASURES:

1. Primary Outcome: Concordance of Genomic Alterations in EGFR Detected in Plasma Versus Tumor Tissue in Stage IV Non Squamous NSCLC Patients Who Are Newly Diagnosed or Progressing on Treatment
Description: Assess concordance of genomic alterations in EGFR detected in plasma (using the OncotypeSEQ Liquid Select assay) versus tumor tissue (assessed centrally using FoundationOne, or locally based on the patient's clinic) in stage IV non squamous NSCLC patients who are newly diagnosed or progressing on treatment.
Time Frame: Time between patient tumor tissue biopsy and and blood collection, up to 8 weeks
Population: Subjects who received EGFR mutation testing on both their tissue and plasma samples.
Measure: Number (95% Confidence Interval); unit: Overall percent agreement (OPA)
Arm/Group | A - NSCLC All Comers Regardless of Genomic Alteration Status
Number analyzed (Participants) | 117
Overall percent agreement (OPA) | 94.0 [88.1 to 97.6]

2. Secondary Outcome: Concordance of Genomic Alterations in ALK (EML4-ALK Fusions) Detected in Plasma Versus Tumor Tissue.
Description: Assess concordance of genomic alterations in ALK (EML4-ALK fusions) detected in plasma (using the OncotypeSEQ Liquid Select assay) versus tumor tissue (assessed centrally using FoundationOne OR locally based on the patient's clinic) in stage IV non squamous NSCLC patients who are newly diagnosed or progressing on treatment.
Time Frame: Time between patient tumor tissue biopsy and and blood collection, up to 8 weeks
Population: Subjects who received ALK (EML4-ALK fusion) mutation testing on both their tissue and plasma samples.
Measure: Number (95% Confidence Interval); unit: Overall percent agreement (OPA)
Groups:
- Patients With Non-squamous NSCLC Either Newly Diagnosed or Pro: Patients with non-squamous NSCLC either newly diagnosed or progressing on any therapy (except erlotinib, gefitinib, or afatinib).
Arm/Group | Patients With Non-squamous NSCLC Either Newly Diagnosed or Pro
Number analyzed (Participants) | 115
Overall percent agreement (OPA) | 95.7 [90.1 to 98.6]

3. Secondary Outcome: Percentage of Participants With EGFR T790M Alterations in Plasma in Patients Progressing on EGFR Targeting Therapy (Erlotinib, Gefitinib, Afatinib).
Description: Detection of EGFR T790M alterations in plasma using the OncotypeSEQ Liquid Select assay. Progression on EGFR targeting therapy (erlotinib, gefitinib, afatinib) assessed clinically or radiologically
Time Frame: Time between patient tumor tissue biopsy and and blood collection (blood collected after the patient progressed on EGFR targeted therapy)
Population: Non-squamous NSCLC patients who progressed on erlotinib, gefitinib, or afatinib treatment and received mutation testing on both their plasma and tissue samples.
Measure: Number; unit: percentage of participants
Groups:
- Patients With Non-squamous NSCLC Who Are Progressing on Erloti: Patients with non-squamous NSCLC who are progressing on erlotinib, gefitinib, or afatinib
Arm/Group | Patients With Non-squamous NSCLC Who Are Progressing on Erloti
Number analyzed (Participants) | 19
percentage of participants | 32

ADVERSE EVENTS:
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Arm/Group | A - NSCLC All Comers Regardless of Genomic Alteration Status | B - Progressing on EGFR Targeted Therapies
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-07): https://cdn.clinicaltrials.gov/large-docs/77/NCT02762877/Prot_SAP_000.pdf